CLINICAL TRIAL: NCT01648842
Title: Vitamin D Status in Pregnant Women With Preeclampsia
Brief Title: Vitamin D and Preeclampsia
Acronym: FEPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: AOM10113
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Vitamin D Deficiency Defined as Serum 25OHD < 75 Nmol/l or 30ng/ml; Preeclampsia; Neonatal Hypercalcemia; Pregnancy
Keywords: Preeclampsia; Vitamin D deficiency; Pregnancy; First trimester
MeSH Terms: conditions — Pre-Eclampsia; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women

SUMMARY:
Hypothesis : Vitamin D serum concentration is decreased in the first trimester in pregnant women who will develop preeclampsia in the second or third trimester compare to a control group Primary purpose : To determine the vitamin D status in the first trimester in a large population of french pregnant women in order to evaluate the importance of the vitamin D deficiency in France and correlate this deficiency with preeclampsia

DETAILED DESCRIPTION:
Primary purpose : To compare the vitamin D (25OHD) status, in the first trimester, in a group of patients with preeclampsia and a group of pregnant women without preeclampsia.

Secondary purpose : (i)To compare the vitamin D status in the third trimester in a group of patients with preeclampsia and a group of pregnant women without preeclampsia. (ii) To evaluate the deficit un vitamin D in a population of pregnant women in the parisian area. (iii) To evaluate the calcemia of the newborns after maternal systematic oral intake of vitamin D 100000U at 28 weeks Methodology : Multicenter (6 centers), Cohort, Nested case-control study Protocol : 4500 patients will be recruited. A blood sample will be performed : in the first trimester (11-14 weeks), in the third trimester (28-40 weeks), and cord blood. For each patient with preeclampsia, 4 controls will be taken from the cohort and matched by parity, race/ethnicity, maternal age, season, BMI. The serum concentration of 25OHD will be measured in all samples.A dosage of 25OHD will be performed in 1000 women from the initial cohort in order to calculate the prevalence of vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* First trimester
* Singleton
* Affiliated to Social security policy
* Woman who gave informed consent

Exclusion Criteria:

* Hypercalcemia (>2.65 mmol/l) or any other phosphocalcic disease
* Hypertension (>140/90) from the first trimester
* Renal insufficiency (creatinine > 120µmol/l)
* Bone disease (osteogenesis imperfecta…)
* Lithium therapy
* Bowel malabsorption
* Kidney stones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Teh vitamin D status will be measured in a large population of french pregnant women (in the first trimester) in order to evaluate the importance of the vitamin D deficency in France and correlate this deficiency with preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 3173 (Actual)
Dates: Start 2012-04-17 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2015-03-16 (Actual)

PRIMARY OUTCOMES:
Vitamin D (25OHD) status in the first trimester | 11-14 (+6) weeks of amenorrhea
  To compare the vitamin D (25OHD) status, in the first trimester, in a group of patients with preeclampsia and a group of pregnant women without preeclampsia

SECONDARY OUTCOMES:
Vitamin D status in the third trimester | 28-40 weeks of amenorrhea
  To compare the vitamin D status in the third trimester in a group of patients with preeclampsia and a group of pregnant women without preeclampsia
Deficit un vitamin D | 11-14 (+6) weeks of amenorrhea
  To evaluate the deficit un vitamin D in a population of pregnant women in the parisian area
Calcemia of the newborns | 1 day (At the moment of the Guthrie test)
  To evaluate the calcemia of the newborns after maternal systematic oral intake of vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra BENACHI, MD/PhD, Principal Investigator — Antoine Béclère Hospital
Locations (1):
- Antoine Béclère Hospital, Clamart, France

REFERENCES:
- [Result] Salakos E, Rabeony T, Courbebaisse M, Taieb J, Tsatsaris V, Guibourdenche J, Senat MV, Haidar H, Jani JC, Barglazan D, Maisonneuve E, Haguet MC, Winer N, Masson D, Elie C, Souberbielle JC, Benachi A. Relationship between vitamin D status in the first trimester of pregnancy and gestational diabetes mellitus - A nested case-control study. Clin Nutr. 2021 Jan;40(1):79-86. doi: 10.1016/j.clnu.2020.04.028. Epub 2020 Apr 25. PMID 32448701